CLINICAL TRIAL: NCT04895189
Title: Yale COVID-19 Recovery Vaccine Study: Measuring Changes in Long Covid Symptoms After Vaccination
Brief Title: Yale COVID-19 Recovery Study
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2000030423; 2U01FD005938-03 (FDA)
Record Dates: First submitted 2021-05-06; First posted 2021-05-20 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Covid19 Sequelae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biospecimen collection will require 45cc of blood and a saliva sample (5 mL) to be given 3 times by each participant. The blood sample will immediately undergo mild agitation and remain stored under controlled temperature. Saliva samples will be self-collected by the participant, who will receive instructions upon arriving at the draw site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention for this observational study. The investigators are observing the changes in participants before and after the participants receive the COVID-19 vaccine, which participants will receive outside of the study.

SUMMARY:
The general purpose of the study is to determine the change in immune responses in people with Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) after vaccination. PASC is a disabling, heterogeneous condition in which people have persistent or emerging symptoms months after an initial SARS-CoV-2 infection, (the virus that causes coronavirus disease 2019, or COVID-19. Specifically, the purpose is to enroll participants suffering from moderate-to-severe PASC prior to vaccination and to measure participants' immune and symptom profiles both before and after vaccination. This study is primarily descriptive.

DETAILED DESCRIPTION:
The investigators are conducting an observational study within Connecticut of adults who have moderate-to-severe PASC and who are planning to receive a vaccine against SARS-CoV-2. The study seeks primarily to describe the heterogeneity in symptoms and immune profile among people with PASC, and once participants have been vaccinated, to determine changes in clinical and immune responses to vaccination and whether there is an association.

Broadly, the study will include 4 surveys to monitor participants' symptom profile and experience with COVID-19 as well as 3 separate biospecimen collection appointments. The surveys and study enrollment will be conducted through REDCap at Yale, a platform that is designed to securely collect survey data from people in a user-friendly design setting. The biospecimen collection will occur at 2 Yale New Haven Health blood draw sites. The biospecimen collection will occur as follows: the first will occur as soon as a participant is enrolled, the second will occur 6 weeks after the participant receives the first dose of a COVID-19 vaccine, and the third will occur 12 weeks after the participant receives the first dose of a COVID-19 vaccine. Participants will be asked to provide 45ccs of blood and a saliva sample (up to 5 mL) for each biospecimen collection. Participants will be able to give a blood sample within a 2-week window (e.g. the collection may be within 5-7 weeks after the participant's first COVID-19 vaccine dose). The survey collection will occur as follows: the first will occur as soon as the participant is enrolled, the second will occur 2 weeks after the participant receives the first dose of a COVID-19 vaccine, the third will occur 6 weeks after the participant receives the first dose of a COVID-19 vaccine, and the fourth will occur 12 weeks after the participant receives the first dose of COVID-19 vaccine. Survey links and reminders will be sent by the Yale research team through REDCap at Yale (via text and/or email) and specimen collection scheduling will be coordinated between the Yale research team and the Yale New Haven Health draw sites.

The study recruitment efforts will be coordinated with YCCI, according to YCCI standards. The investigators will also distribute a study flyer at local Long Covid health clinics and on social media, including Twitter and Facebook. In addition to recruitment efforts at Yale, the investigators' patient partners, Survivor Corps, will be publicizing the study by sharing the study information and eligibility requirements on social media including Facebook and Twitter. Survivor Corps's recruitment efforts will not be coordinated by the Yale research team. There will be a study landing page where potential participants can find information about the study and the study link.

Potential participants will be provided a link for the study enrollment as well as an email address (covidrecovery@yale.edu) to reach out for more information about the study. The study enrollment process will take place on REDCap at Yale and by phone. Participants will complete a brief screening questionnaire to determine study eligibility and to provide an email address and/or phone number. Study coordinators will then reach out, by email to schedule a phone consultation, or directly by phone, as is the participant's preference. During the phone consultation, a study coordinator will read a script designed to inform the participant of the study design and risks to ensure that the participant understands the study prior to consent. The participant will also be asked if the participant has any questions for the study coordinator. Once the phone consultation is complete, the study coordinator will email the participant a link to the e-consent, which will be a REDCap form. Once the participant consents to the study, which will require an e-signature, a study coordinator will sign a REDCap form to acknowledge that the e-consent is complete. An email will automatically be sent to the participant containing the (REDCap) link for the first survey and information as to how to provide the first biospecimen sample. The research team will also contact the participant within the next 2-3 days by phone to provide information regarding the timing and location for biospecimen collection and to answer any questions the participant has.

Participants will provide blood and saliva samples 3 times at any of the study's 2 Yale New Haven Health blood draw sites. While all specimen collection will occur in Connecticut at these sites, people who are not currently patients within the Yale New Haven Health system will still be eligible to participate in the study, so long as the participant is willing and able to travel to one of the blood draw sites 3 times. The Yale study consent will include consenting to providing blood and saliva samples 3 times at a Yale New Haven Health site.

This research will foster a community spirit with participants, producing a collaboration based on relationships, not merely transactions. The Survivor Corps group has joined this effort and will ensure that the study includes the participant perspective and abide by the study's principles. Survivor Corps is an independent group of people who experienced long-term effects of SARS-CoV-2 infection and seek to generate knowledge about people with prolonged recoveries. The Patient-Led Research Collaborative has also joined this effort to provide a PASC participant perspective on the study's participant-facing communication and surveys. Patient-Led Research is also an independent group of people who experienced long-term effects of SARS-CoV-2 infection and seek to generate knowledge about people with prolonged recoveries.

The study will utilize REDCap at Yale to screen for eligibility, conduct e-consent, and to collect survey information. The data will reside within the secure platform and will be transferred to Yale via a secure file transfer service. The data will then reside on secure servers at Yale.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English or Spanish
2. Age 18 years and over
3. Test positive for SARS-CoV-2 (defined as a patient who reports receiving any screening or diagnostic test used to detect the presence of SARS-CoV-2 including any FDA-approved or authorized molecular or antigen-based assay) at least 2 months prior to the start of this study OR test positive for antibodies to SARS-CoV-2 at any point OR receive a positive T-test at any point OR receive a clinical diagnoses of COVID-19 at any point OR was hospitalized due to COVID-19 at any point
4. Self-report moderate to severe symptoms or disability due to PASC
5. Self-report planning to receive a vaccine against SARS-CoV-2
6. Self-report has not yet received any doses of a vaccine against SARS-CoV-2

Exclusion Criteria:

1. Unable to provide informed consent
2. Unable to provide 3 blood and saliva samples at one of the 2 participating Yale New Haven Health blood draw sites on a Monday or Wednesday morning (before 12 pm).
3. Does not have access to a hand-held device or computer that would allow for digital participation in the study
4. Do not have and do not want to set up an email address
5. Individuals who are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will include adults aged 18 and over who either have been diagnosed with COVID-19, hospitalized due to COVID-19, or who have tested positive for SARS-CoV-2 more than 2 months prior to joining the study (PCR, antigen, or a positive T-test or antibody test at any point), and who have proof of the diagnosis, hospitalization, or positive test; who intend to receive the vaccine for SARS-CoV-2, but who have not yet received any doses of the vaccine; and who self report having persistent moderate-to-severe symptoms or disability.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Surveys 2-4 Effect of Vaccination | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  The primary outcome for the study is whether people's overall health condition improves, does not change, or worsens after receiving the COVID-19 vaccine. This outcome will be measured with the question in Surveys 2-4: "Would you say that your overall health, as compared to your health before the vaccine, is worse, better, or the same?" The number of participants within each group will be reported.
Immune Assay Findings | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  For each group of participants by overall health condition change, immune response trends that were found through saliva-based or blood-based analyses will be reported. Trends found in the immune cells, antibodies, and viral loads of participants for whom symptoms either improved, worsened, or did not change after vaccination will be reported.

SECONDARY OUTCOMES:
Surveys 1-4 Overall Change in Symptoms | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  The symptoms, as identified in Survey 1, will be measured across the study period and the overall change will be captured by Surveys 2-4. The study outcome will be reported by both symptom clusters and individual symptoms. Overall symptom change will be described by whether participants report that symptoms have improved, changed, or stayed the same since before the vaccine. Symptom clusters will be data-driven; symptoms will not be grouped based on pre-specified categories.
Surveys 2-4 Change in Symptom Severity | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  The symptoms, as identified in Survey 1, will be measured across the study period and the change in symptom severity will be captured by Surveys 2-4. The study outcome will be reported by both symptom clusters and individual symptoms. The change in symptom severity will be described by whether participants report that symptoms have become more severe, less severe, or did not change severity since before the vaccine. Symptom clusters will be data-driven; symptoms will not be grouped based on pre-specified categories.
Surveys 2-4 Change in Symptom Frequency | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  The symptoms, as identified in Survey 1, will be measured across the study period and the change in symptom frequency will be captured by Surveys 2-4. The study outcome will be reported by both symptom clusters and individual symptoms. The change in symptom frequency will be described by whether participants report that symptoms have become more frequent, less frequent, or did not change in frequency since before the vaccine. Symptom clusters will be data-driven; symptoms will not be grouped based on pre-specified categories.
Surveys 2-4 Change in Symptom Duration | The measure will be reported both longitudinally, over the 3 months following the participant post-vaccination (reporting the result at 2 weeks, 6 weeks, and 12 weeks post-vaccination), and as a cross-sectional result at the end of the study (week 12).
  The symptoms, as identified in Survey 1, will be measured across the study period and the change in symptom duration will be captured by Surveys 2-4. The study outcome will be reported by both symptom clusters and individual symptoms. The change in symptom duration will be described by whether participants report that symptoms have lasted for more, less, or the same amount of time since before the vaccine. Symptom clusters will be data-driven; symptoms will not be grouped based on pre-specified categories.

CONTACTS AND LOCATIONS:
Overall Officials: Harlan Krumholz, MD, SM, Principal Investigator — Director, Center for Outcomes Research and Evaluation (CORE)
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Study investigators may share aggregate and deidentified data with other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will become available once data collection is complete, in approximately May of 2022. The data will be deleted after 10 years.

REFERENCES:
- [Result] Grady CB, Bhattacharjee B, Silva J, Jaycox J, Lee LW, Silva Monteiro V, Sawano M, Massey D, Caraballo C, Gehlhausen JR, Tabachnikova A, Mao T, Lucas C, Pena-Hernandez MA, Xu L, Tzeng TJ, Takahashi T, Herrin J, Guthe DB, Akrami A, Assaf G, Davis H, Harris K, McCorkell L, Schulz WL, Griffin D, Wei H, Ring AM, Guan L, Dela Cruz C, Krumholz HM, Iwasaki A. Impact of COVID-19 vaccination on symptoms and immune phenotypes in vaccine-naive individuals with Long COVID. Commun Med (Lond). 2025 May 9;5(1):163. doi: 10.1038/s43856-025-00829-3. PMID 40346201